CLINICAL TRIAL: NCT03646890
Title: Epidemiology and Clinical Features of Uveitis in a Tertiary Referral Center in Montpellier, France
Brief Title: Epidemiology and Clinical Features of Uveitis in a Tertiary Referral
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0280
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Uveitis
Keywords: Epidemiology; Clinical features; Etiology; Tertiary center
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to report the pattern of uveitis in patients attending a tertiary referral center at the University hospital in Montpellier. The patients seen at the specialized consultation for uveitis between 2002 and first semester 2018 were included.

Data about demography, clinical features and final diagnoses were collected and updated during the differenet visits. The medical records were restrospectively rewieved and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen at the specialized consultation for uveitis between 2002 and first semester 2018

Exclusion Criteria:

* Patients under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at the specialized consultation for uveitis between January 2002 and july 2018
Sampling Method: Non-Probability Sample
Enrollment: 985 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2012-01-01 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Etiology of uveitis | 1 day
  Etiology of uveitis

SECONDARY OUTCOMES:
Demographic description of patients with uveitis | 1 day
  Demographic description of patients with uveitis
Clinical description of patients with uveitis | 1 day
  Clinical description of patients with uveitis

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Schneider, PUPH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC